CLINICAL TRIAL: NCT00367965
Title: The Effect of Eszopiclone 3 mg Compared to Placebo on Daytime Function in Subjects With Insomnia Related to Rheumatoid Arthritis
Brief Title: Study of Eszopiclone Compared to Placebo on Daytime Function in Subjects With Insomnia Related to Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-055
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia; Arthritis, Rheumatoid
Keywords: Insomnia related to rheumatoid arthritis (RA)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Arthritis, Rheumatoid | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): eszopiclone 3 mg
  Interventions: Drug: Eszopiclone
- 2 (Placebo Comparator): placebo tablet
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Eszopiclone — eszopiclone 3 mg
  Other Names: Lunesta; S-zopiclone
  Arms: 1
Drug: placebo — placebo tablet
  Arms: 2

SUMMARY:
To demonstrate subjective sleep efficacy of eszopiclone 3 mg in subjects with insomnia related to rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind, placebo controlled, parallel group study of eszopiclone 3 mg in subjects with insomnia related to rheumatoid arthritis. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Subject must understand the purpose of the study and be willing to adhere to the study schedule and procedures described in this protocol.
* Subject must be 25-64 years of age (inclusive) on the day of signing consent.
* Subject must be diagnosed with rheumatoid arthritis as defined by the American College of Rheumatology.
* Subject must be on stable regimen for treatment of rheumatoid arthritis for a minimum of 90 days prior to study start.
* Subject must report a wake time after sleep onset (WASO) of greater than or equal to 45 minutes and less than or equal to 6.5 hours of total sleep time at least three times a week over the previous month and symptoms of insomnia must post date onset of rheumatoid arthritis.
* Subject physical exam must show no clinically significant abnormal findings (other than those related to rheumatoid arthritis) at screening.
* Subject must have no clinically significant abnormal laboratory findings at screening (other than those related to rheumatoid arthritis).
* Subject must have no clinically significant ECG abnormalities at screening.

Exclusion Criteria

* Subject has diagnosis of fibromyalgia, or juvenile rheumatoid arthritis.
* Subject has history of circadian rhythm disorder, or travels across >3 time zones on a regular basis.
* Female subject is pregnant, lactating or within 6-months post partum.
* Subject has a history of drug or alcohol abuse or dependence in the past 2 years or positive urine drug test at screening.
* Subject has clinically significant unstable medical abnormality or unstable chronic disease (other than insomnia and rheumatoid arthritis) including severe cardiac, renal, or hepatic or respiratory disease, seizure disorder.
* Subject has participated in any investigational drug study within 30 days prior to screening or plans to participate in any investigational drug study during participation in this study.
* Subject has a history of malignancy within 5 years, or current malignancy, except for non-melanoma skin cancer.
* Subject has a current primary psychiatric diagnosis of any of the following disorders: dementia, delirium, schizophrenia, psychosis, other psychotic disorders, dysthymic disorder; major depressive disorder, bipolar disorders; cyclothymic disorder, other mood disorders, primary anxiety disorders, primary panic disorders, or any nocturnal panic disorder.
* Subject has any of the following Personality Disorders diagnoses: schizotypal, schizoid, borderline personality disorder; or any other personality disorder that would compromise the investigator's ability to evaluate the safety and efficacy of the study medication.
* Subject has difficulties in sleep initiation or maintenance associated with known medical diagnosis [e.g. sleep apnea]; diagnosed and untreated restless leg syndrome (RLS) or periodic leg movement syndrome (PLMS).
* Subject has used any drugs known or suspected to affect hepatic or renal clearance capacity within a period of 30 days prior to screening.
* Subject reports consumption of more than two alcoholic beverages daily, 14 or more alcoholic beverages weekly, or five or more alcoholic beverages on any given day.
* Subject is a rotating or third/night shift worker.
* Subject is a staff member or relative of a staff member.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2004-02; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
mean subjective wake time after sleep onset (WASO) | Week 1

SECONDARY OUTCOMES:
WASO | Weeks 2, 3, and 4
Number of nocturnal awakening | Weeks 1, 2, 3, and 4
Total sleep time (TST) | Weeks 1, 2, 3, and 4
Sleep Efficiency | Weeks 1, 2, 3, and 4
Sleep latency (SL) in subjects with sleep latency of 30 minutes or greater at screening | Weeks 1, 2, 3, and 4
Quality of sleep | Weeks 1, 2, 3, and 4
Depth of sleep | Weeks 1, 2, 3, and 4
Daytime alertness | Weeks 1, 2, 3, and 4
Ability to concentrate | Weeks 1, 2, 3, and 4
Physical well-being | Weeks 1, 2, 3, and 4
Ability to function | Weeks 1, 2, 3, and 4
occurrence of rebound insomnia and withdrawal effects will be assessed for WASO, and TST as well as for SL in subjects with sleep latency of 30 minutes or greater at screening | Weeks 1, 2, 3, and 4
Duration of morning stiffness | Weeks 1, 2, 3, and 4
Pain severity (from IVRS) | Weeks 1, 2, 3, and 4
Epworth Sleepiness Scale | Weeks 2 and 4
Insomnia Severity Index | Weeks 2 and 4
Arthritis Self-Efficacy Scale | Week 4
SF-36 | Week 4
Physician Clinical Global Impression of treatment | Week 4
ACR Response Criteria | Week 4
Percentage of subjects with increase in dose or new prescription of pain medications | Weeks 1, 2, 3, 4
Percentage of subjects with increase in dose or new prescription of disease modifying medications | Weeks 1, 2, 3, 4

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Huntsville, Alabama
  - Tucson, Arizona
  - Santa Maria, California
  - Whittier, California
  - Danbury, Connecticut
  - Hamden, Connecticut
  - Washington D.C., District of Columbia
  - Aventura, Florida
  - Clearwater, Florida
  - Fort Lauderdale, Florida
  - Ocala, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Springfield, Illinois
  - Kansas City, Kansas
  - Overland Park, Kansas
  - Louisville, Kentucky
  - Fall River, Massachusetts
  - Lansing, Michigan
  - St Louis, Missouri
  - Medford, New Jersey
  - Rochester, New York
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Mayfield Village, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Bethlehem, Pennsylvania
  - Norristown, Pennsylvania
  - West Reading, Pennsylvania
  - Columbia, South Carolina
  - Myrtle Beach, South Carolina
  - Memphis, Tennessee
  - Amarillo, Texas
  - Dallas, Texas
  - Lubbock, Texas
  - Everett, Washington

REFERENCES:
- [Derived] Roth T, Price JM, Amato DA, Rubens RP, Roach JM, Schnitzer TJ. The effect of eszopiclone in patients with insomnia and coexisting rheumatoid arthritis: a pilot study. Prim Care Companion J Clin Psychiatry. 2009;11(6):292-301. doi: 10.4088/PCC.08m00749bro. PMID 20098520